CLINICAL TRIAL: NCT00387647
Title: A Multicenter, Phase 2 Study of Maintenance Azacitidine in Elderly Patients With Acute Myeloid Leukemia in Complete Remission After Induction Chemotherapy
Brief Title: Maintenance Azacitidine in Elderly Patients With Acute Myeloid Leukemia (AML) in CR After Induction Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14496; NCT00365664 (obsolete NCT alias)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia
Keywords: myeloid; acute; monocytic
MeSH Terms: conditions — Leukemia | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine Treatment (Experimental): Azacitidine 50 mg/m^2 subcutaneously daily for 5 days (Monday through Friday) on days 1 through 5, every 28 days for 6-12 cycles.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine given subcutaneously as outlined in treatment arm.
  Other Names: Vidaza™

SUMMARY:
The purpose of this study is to find out if patients older than 60, with acute myeloid leukemia, who are in complete remission following initial chemotherapy, will live longer and have a lower rate of leukemia relapse when treated with azacitidine.

DETAILED DESCRIPTION:
Patient activity will encompass approximately 48 months: an approximate 24 month enrollment period, followed by 6 to 12 months of patient treatment. Patients will be followed for 1 year following completion of study drug treatment. During follow-up, bone marrow biopsies to confirm disease status should be obtained if peripheral blood blasts are present or if there is development of unexpected blood abnormalities to warrant suspicion of relapse, or at a minimum of every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of AML with greater than 20% blasts in bone marrow. All AML subtypes of the World Health Organization (WHO) classification will be included with the exception of promyelocytic leukemia and cytogenetics showing the (15;17) translocation or AML secondary to chemotherapy.
* Achieved first morphologic complete remission (CR) or first morphologic complete remission with incomplete platelet recovery (CRp) after completion of induction chemotherapy using a standard induction regimen. Up to 2 induction cycles will be allowed. Confirmation of CR is defined as < 5% blasts in the bone marrow specimen, with a count of at least 100-200 nucleated cells and absence of Auer rods, along with peripheral blood neutrophil count >1.0 x 10^9/L and platelet count >100 x 10^9/L. Confirmation of CRp is defined as <5% blasts in the bone marrow specimen, with a count of at least 100-200 nucleated cells and absence of Auer rods, with incomplete platelet recovery (ANC ≥ 1000/µL and platelets 50-99,000/µL, along with transfusion-independence of red blood cells).
* Received up to 2 cycles of any consolidation chemotherapy
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Normal organ function at the time of screening: Total bilirubin ≤1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN; Serum creatinine ≤1.5 x ULN or creatinine clearance >60 mL/min for patients with creatinine levels above ULN
* Men must agree to avoid fathering a child throughout the study.
* Be capable of giving informed consent and have signed the informed consent form (ICF)

Exclusion Criteria:

* Greater than 12 weeks since initiation of most recent cycle of consolidation chemotherapy
* Women of childbearing potential
* Prior relapse after complete remission for AML
* AML secondary to previous exposure to cytotoxic chemotherapy known to induce leukemia
* Active malignancy other than AML
* Any diagnosis of metastatic disease
* Have hepatic tumors
* Radiation therapy, chemotherapy, or cytotoxic therapy, given to treat conditions other than AML <4 weeks prior to Day 1 or have not recovered from adverse events due to agents administered >4 weeks earlier
* Known leukemic involvement of the central nervous system
* Known or suspected hypersensitivity to azacitidine or mannitol
* Prior or active disease that, in the opinion of the Investigator, may interfere with the procedures or evaluations to be conducted in the study (uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements)
* Active viral infection with known human immunodeficiency virus (HIV) or viral hepatitis type B or C
* Treatment with other investigational drugs within the 30 days prior to Day 1, or ongoing adverse events from previous treatment with investigational drugs, regardless of the time period
* Any prior treatment with azacitidine or decitabine

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-08; Primary Completion 2013-10 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Lancet, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Researchers consented 29 potential participants between 08/02/0206 and 11/01/2011. 24 eligible participants began treatment, one at Duke University Medical Center and 23 at Moffitt Cancer Center.
Groups:
- Azacitidine Treatment: Azacitidine 50 mg/m^2 subcutaneously daily for 5 days (Monday through Friday) on days 1 through 5, every 28 days for 6-12 cycles. Patients were to be followed for 1 year following completion of study drug treatment.
Period: Overall Study
Arm/Group | Azacitidine Treatment
Started | 24
Completed | 6
Not Completed | 18
Not completed — Death | 18

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Azacitidine Treatment
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 68.7 [62 to 81]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Rate of Disease Free Survival at One Year
Description: The primary efficacy variable is disease free survival measured at one year, which is the percentage of patients who remain alive and disease free one year after the confirmation of remission by bone marrow biopsy. Relapse is defined by a bone marrow specimen with >5% blasts or the presence of Auer rods.
Time Frame: 1 year
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine Treatment
Number analyzed (Participants) | 24
percentage of participants | 50 [lower limit 7.3]

2. Secondary Outcome: Overall Survival (OS)
Description: The secondary efficacy variable is overall survival measured as time to death, which is the time from remission until death from any cause.
Time Frame: 48 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine Treatment
Number analyzed (Participants) | 24
months | 20.4 [12.2 to 26.0]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety and tolerability of treatment as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Time Frame: 48 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Azacitidine Treatment
Number analyzed (Participants) | 24
participants | 24

ADVERSE EVENTS:
Time Frame: 6 years, 1 month overall
Description: Adverse event observation from after study drug administration on cycle 1 /day 1, through 28 days following the last dose of azacitidine.
Arm/Group | Azacitidine Treatment
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine Treatment (N=24)
Colitis, infectious (e.g., Clostridium difficile) - possibly related (Infections and infestations) | 1 (1)
Dyspnea (shortness of breath), unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine Treatment (N=24)
Platelets - low (Blood and lymphatic system disorders) | 19 (81)
Neutrophils/granulocytes (ANC/AGC) - low (Blood and lymphatic system disorders) | 18 (73)
Leukocytes (total WBC) - low (Blood and lymphatic system disorders) | 15 (57)
Hemoglobin - low (Blood and lymphatic system disorders) | 3 (9)
Constipation (Gastrointestinal disorders) | 11 (20)
Nausea (Gastrointestinal disorders) | 7 (7)
Anorexia (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 10 (23)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (11)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3 (11)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Pain - Head/headache (General disorders) | 4 (7)
Pain - Abdomen NOS (General disorders) | 3 (4)
Pain - Back (General disorders) | 2 (2)
Pain - Dental/teeth/peridontal (General disorders) | 2 (2)
Pain - Extremity-limb (General disorders) | 2 (2)
Pain - Other (General disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (11)
Constitutional Symptoms - Other (General disorders) | 2 (2)
Fever (in the absence of neutropenia) (General disorders) | 2 (4)
Sweating (diaphoresis) (General disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 6 (8)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3 (3)
Ocular/Visual - Other (Eye disorders) | 4 (4)
Hypotension (Cardiac disorders) | 2 (3)
Auditory/Ear - Other (Ear and labyrinth disorders) | 2 (3)
Cardiac Arrhythmia - Other (Cardiac disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Only five participants completed study and defined follow-up period and one participant remained on follow-up at time of analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes